CLINICAL TRIAL: NCT05862727
Title: Preschool Attention and Sleep Support (PASS): A Telehealth Intervention for Children at Risk for ADHD
Brief Title: Preschool Attention and Sleep Support (PASS)
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00111845; R34MH131994-01 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-05-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Psychiatric Health
Keywords: Psychiatric Health; Children; Preschool; ADHD; Telehealth Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Behavioral Telehealth Intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to one of two interventions, and will not be told which intervention they are assigned to. Outcomes assessor will also be blinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASS Arm1 (Experimental): Caregivers will receive sessions of evidence-based behavioral parent training which focuses on improving behaviors, such as establishing daytime and bedtime routines, through enhancement of positive parenting skills, including modifying antecedents, applying/withdrawing positive attention as a consequence, and shaping behavior using salient rewards.
  Interventions: Behavioral: Telehealth Intervention
- PASS Arm2 (Active Comparator): Caregivers will receive sessions of evidence-based behavioral parent training which focuses on improving behaviors, including in home and public settings, through enhancement of positive parenting skills, including modifying antecedents, applying/withdrawing positive attention as a consequence, and shaping behavior using salient rewards.
  Interventions: Behavioral: Telehealth Intervention

INTERVENTIONS:
Behavioral: Telehealth Intervention — Telehealth intervention that teaches caregivers evidence-based skills and provides practice opportunities to manage their children's ADHD-related behaviors according to their assigned intervention.

SUMMARY:
This study will be investigating two telehealth interventions for preschoolers with ADHD. The study is divided into two Aims. During Aim 1, caregivers of preschoolers with attention concerns, pediatric behavioral health professionals, and pediatric primary care providers will take part in two virtual focus groups to provide their perspective on ways to improve the telehealth intervention being evaluated.

DETAILED DESCRIPTION:
During Aim 2, caregivers of preschool children with ADHD symptoms will be randomly assigned to participate in one of two 9-week telehealth interventions. Both interventions will teach evidence-based skills and provide practice opportunities to manage their children's ADHD-related behaviors. Caregivers and their children will also attend three study visits (one before the intervention, and two following the intervention) where they will be asked to complete questionnaires and assessments related to the child's ADHD symptoms, psychiatric health, and sleep habits. Following each study visit, participating children will be asked to wear an ActiGraph device on their nondominant wrist for 24 hours/day for a 7-day period. During this time, the caregivers will be asked to complete an electronic daily diary about their child's sleep.

ELIGIBILITY:
Inclusion Criteria:

* child must be ages 3-5 years at intake
* child with score of 30 on the Child Sleep Habits Survey-Short Form and a caregiver rating of child's sleep problems as moderate/severe
* child with ≥80th percentile on the clinician-rated ADHD-RS based on age and sex norms, with at least 4 symptoms in the clinically significant range (scores of 2-3) in either the inattention or hyperactive/impulsive domains
* parent/caregiver must have ability to speak, read, and write in English
* parent/caregiver must have access to a device with internet and/or smartphone to access telehealth visits
* parent/caregiver must have ability to follow written and verbal instructions
* parent/caregiver must have ability and willingness to comply with study procedures.

Exclusion Criteria:

* child with suspected obstructive sleep apnea or restless legs syndrome (via screening questionnaires)
* child with current use of stimulant medication, other psychotropics, or medications for sleep (prescription or over-the-counter, including melatonin)
* child with caregiver report of psychiatric disorder other than ADHD requiring treatment (medication and/or therapy), Autism Spectrum Disorder, or intellectual disability
* parent/caregiver is currently participating in another parent training intervention or have previously participated in another parent training intervention in the past 6 months.
* Severe and/or uncontrolled medical condition (e.g., pulmonary and neurological conditions such as cystic fibrosis and seizure disorder) that would interfere with sleep and/or study participation according to the study team

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Change in clinician-rated ADHD-RS | Baseline, immediately post-treatment, 3 months post-treatment
  A clinician-rated, 18-item assessment with a 4-point Likert scale ranging from Rarely or never to Very Often.
  Lower scores indicate better outcomes.
Change in caregiver-reported sleep habits as measured by the Short-Form Child Sleep Habits Questionnaire (SF-CSHQ). | Baseline, immediately post-treatment, 3 months post-treatment
  A 23-item questionnaire with a 3-point Likert scale ranging from Rarely to Usually. Lower scores indicate better outcomes.
Change in Sleep Regularity Index (SRI) | Baseline, immediately post-treatment, 3 months post-treatment
  A measure of sleep regularity collected continuously over 7 days via Actigraphy. The SRI is calculated as the proportion of pairs of time points 24 hours apart that have matching sleep/wake status

SECONDARY OUTCOMES:
Change in psychosocial function as measured by Impairment Rating Scale | Baseline, immediately post-treatment, 3 months post-treatment
  A clinician rated, 8-item assessment with a 7-point Likert scale ranging from No problem; definitely does not need treatment/special services to Extreme Problem; definitely needs treatment/special services. Lower scores indicate better outcomes.
Change in parenting stress as measured by the Parenting Stress Scale | Baseline, immediately post-treatment, 3 months post-treatment
  An 18-item questionnaire with a 5-point Likert Scale ranging from Strongly disagree to Strongly Agree. Lower scores indicate better outcomes.
Change in comorbid symptoms as measured by Child Behavioral Checklist for Ages 1½ to 5(CBCL) | Baseline, immediately post-treatment, 3 months post-treatment
  A widely-used 99-item parent report questionnaire with a 3-point Likert Scale ranging from Not True to Very True or Often True. Lower scores indicate better outcomes.
Change in sleep midpoint, TST (minutes from sleep start to sleep end), SOL (minutes to first sleep epoch), WASO (minutes awake between sleep start and sleep end), and SE (TST/time in bed). | Baseline, immediately post-treatment, 3 months post-treatment
  As measured via actigraphy collected continuously over 7 days.
Change in parenting style as measured by the Alabama Parenting Questionnaire | Baseline, immediately post-treatment, 3 months post-treatment
  A 33-item questionnaire with a 5-point Likert Scale ranging from Never to Always.
Change in severity of behavior problems in the home setting as measured by the Home Situations Questionnaires. | Baseline, immediately post-treatment, 3 months post-treatment
  A 16-item questionnaire with a 9-point Likert Scale. Lower scores indicate better outcomes.

OTHER OUTCOMES:
Treatment Fidelity | During the 9-week treatment
  The percentage of content and practices of the PASS protocol that were delivered (yes/no) across providers as determined by rater's assessment of recorded sessions.
Feasibility of Recruitment | Baseline
  The percentage of enrolled participants who attend a screening visit.
Feasibility of Randomization | Baseline
  The percent of randomized participants who meet study eligibility after attending the screening visit.
Integrity of the control condition as measured by the PASS Fidelity Checklist. | During the 9-week treatment
  The incidence of administration of core PASS elements in each session of the control group determined by rater.
Integrity of the control condition as measured by the Integrity of the Blind questionnaire. | immediately post-treatment
  Asking all blinded informant (parents, assessors) to guess whether the child was in the control or experimental group and to state their confidence in this guess on a 1 to 10 scale. Higher scores indicate higher confidence in guess.
Index of treatment engagement as measured by attendance. | During the 9-week treatment
  Average number PASS groups sessions attended by participants.
Adherence to between-session practice. | During the 9-week treatment
  Assessed via a therapist-completed item assessing the degree to which the caregiver was adherent overall with homework immediately after each session on a scale of 1 (not at all) to 5 (extremely strong).
Retention | Immediately post-treatment, 3 months post-treatment
  Measured by the number of families who complete post-treatment and follow-up assessments.
Acceptability as measured by the Satisfaction with Therapy and Therapist Scale (STTS-R). | Immediately post-treatment
  A 13-item questionnaire with a 5-point Likert Scale ranging from Strongly Disagree (1) to Strongly Agree (5). Higher scores indicate better outcomes.
The Client Credibility Questionnaire | Immediately post-treatment
  4 item questionnaire to determine how logical and successful the treatment is; if they would recommend the intervention to others; and how much symptoms improved.
Parenting Sense of Competence Scale | Baseline, immediately post-treatment, 3 months post-treatment
  A 17-item questionnaire with a 6-point Likert Scale ranging from Strongly Disagree (1) to Strongly Agree (6). A higher score indicates a higher parenting sense of competency.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lunsford-Avery, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial (including data dictionaries) will be available for this study after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be accessible by researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals and questions for data access should be directed to NDAHelp@mail.nih.gov. To gain access, data requestors will need to sign a data access agreement at https://nda.nih.gov/nda/access-data-info.html.
URL: https://nda.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT05862727/ICF_000.pdf